CLINICAL TRIAL: NCT04485637
Title: Helping Hypertension Patients to Interpret Blood Pressure Readings and Motivate Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Wandi Bruine de Bruin, Provost Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BloodPressureCommunications
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Communication with basic table (Other): Blood pressure communication showing a basic table representing only the normal range of blood pressure readings
  Interventions: Other: Communication with basic table
- Communication with enhanced table (Other): Communication showing an enhanced table (Fig 1B) with more reference information for interpreting blood pressure readings, including how combinations of diastolic and systolic blood pressure reflect normal, elevated and hypertension ranges (adapted from the American Heart Association)
  Interventions: Other: Communication with enhanced table
- Communication with enhanced graph (Other): Communication showing an enhanced graph (adapted from Blood Pressure UK) for interpreting blood pressure readings, showing the same color-coded ranges as the enhanced table, with diastolic blood pressure on the x-axis and systolic blood pressure on the y-axis
  Interventions: Other: Communication with enhanced graph

INTERVENTIONS:
Other: Communication with basic table — Communication showing only the normal range of blood pressure readings, which is often used but may make it hard to interpret numbers outside of the normal range
  Arms: Communication with basic table
Other: Communication with enhanced table — Communication with enhanced table, with reference information showing how combinations of diastolic and systolic blood pressure reflect normal, elevated and hypertension ranges (adapted from the American Heart Association)
  Arms: Communication with enhanced table
Other: Communication with enhanced graph — Communication with enhanced graph, showing reference information about how to interpret blood pressure readings (adapted from Blood Pressure UK) with diastolic blood pressure on the x-axis and systolic blood pressure on the y-axis
  Arms: Communication with enhanced graph

SUMMARY:
Hypertension is a major risk factor for cardiovascular disease, and a leading cause of death worldwide. Only about 50% of hypertension patients have good blood pressure control, perhaps because they find it hard to understand their blood pressure readings. The investigators will evaluate ways to help hypertension patients to interpret their blood pressure readings and motivate blood pressure control.

Aim 1: Based on existing communications, the investigators will create 3 blood pressure communications:

(A) a basic table showing only the normal blood pressure range, which is often used in clinical practice and online communications about blood pressure, but may make it hard to interpret numbers outside of the normal range, potentially undermining behavior change intentions; (B) an enhanced table showing how combinations of diastolic and systolic blood pressure reflect normal, elevated and hypertension ranges, from the American Heart Association; (C) an enhanced graph to be adapted from Blood Pressure UK to show the same color-coded ranges as the enhanced table, with diastolic blood pressure on the x-axis and systolic blood pressure on the y-axis.

Aim 2: : Among 650 diagnosed hypertension patients recruited through the University of Pittsburgh Medical Center (UPMC) Pitt+Me Patient Registry, the investigators will evaluate whether being presented with the enhanced table or graph (vs. basic table) affects patients' self-reported blood pressure measurement (as averaged across two measurements taken at the time of the survey at least 1 minute apart, as per directions of the American Heart Association), and improves interpretations of these two blood pressure readings and of hypothetical blood pressure readings, as well as behavior change intentions.

Aim 3: The investigators will examine whether Aim 2 findings vary by health literacy, age, and SES.

DETAILED DESCRIPTION:
BACKGROUND Hypertension is a major modifiable risk factor for cardiovascular disease, and a leading cause of death worldwide. Lifetime risk of hypertension is 70-90%, but it is higher among adults who are older and of low socio-economic status (SES). Older age and lower SES are also associated with low health literacy, which undermines understanding of health information. Yet, low health literacy in hypertension patients is an independent predictor of poor blood pressure control, with only about 50% of hypertension patients having controlled blood pressure. Possibly, patients with lower health literacy find it harder to interpret whether blood pressure readings are high or low, reflect good or bad blood pressure control, and indicate a need for behavior change or medication use. Even college-educated hypertension patients who have bought home blood pressure monitors may struggle to interpret blood pressure readings that are outside the normal range, undermining their intentions to improve their blood pressure control.

BEHAVIORAL SCIENCE INSIGHT Lab studies in behavioral science have found that individuals' ability to interpret numbers (likely including blood pressure readings) is improved by showing the range or distribution - also called 'reference information'. In preliminary work, the PI showed that many people struggle to interpret credit card APRs, because they do not know what numbers are good or bad. In line with the behavioral science insight, the PI found that providing graphs with ranges of existing APRs helped recipients to see which credit cards posed a bad deal, and reduced their intentions to get such credit cards. It has been posited that providing reference information (e.g. normal and abnormal blood pressure ranges) should also help hypertension patients to interpret blood pressure readings, and help them to control their blood pressure.

If reference information is used when communicating blood pressure readings in clinics and online health records, it often involves a basic table that only shows the normal range (e.g., <120 for systolic and <80 for diastolic blood pressure). In one behavioral science study, 106 university staff performed similarly when using this basic table or when using a color-coded horizontal bar graph (showing the normal range in white and values outside the normal range in black). However, neither format followed the American Heart Association's communication, which shows more reference information for interpreting blood pressure readings outside of the normal range. Hypertension patients may need to see such enhanced reference information, because they are more likely to encounter blood pressure readings outside of the normal range. Moreover, those readings can be harder to interpret - perhaps especially for hypertension patients with low health literacy. The investigators propose to evaluate 2 formats for providing the more enhanced reference information from the American Heart Association, in either a table (as used by the American Heart Association), or a graph (as used by Blood Pressure UK, to be adapted to show the information from the American Heart Association). The behavioral science literature suggests that tables facilitate reading specific numbers, but that graphs help more with interpreting numbers as high or low, and good or bad - though that could depend on recipients' health literacy.

SPECIFIC AIMS The American Heart Association has called for broad-based efforts to improve the proportion of hypertension patients with controlled blood pressure, by "further engaging individuals in the hypertension control process" with "adequate representation of [specific] populations" including those with lower health literacy, older age, and lower SES. Therefore, the investigators propose to conduct an NIH Stage I primary data collection project, to evaluate the efficacy of interventions to facilitate blood pressure readings and motivate blood pressure control, in a sample of hypertension patients varying in health literacy, age, and SES.

Aim 1: Based on existing communications, the investigators' communication expertise (see below), and pilot tests with up to 10 hypertension patients, the investigators will generate 3 blood pressure communications:

(A) a basic table showing only the normal range, which is often used but may make it hard to interpret numbers outside of the normal range, potentially undermining behavior change intentions; (B) an enhanced table with more reference information, showing how combinations of diastolic and systolic blood pressure reflect normal, elevated and hypertension ranges, from the American Heart Association; (C) an enhanced graph to be adapted from Blood Pressure UK to show the same color-coded ranges as the enhanced table, with diastolic blood pressure on the x-axis and systolic blood pressure on the y-axis.

Aim 2:: In a sample of 650 diagnosed hypertension patients recruited through the Pitt+Me Patient Registry at the University of Pittsburgh Medical Center (UPMC), the investigators will evaluate whether being presented with the enhanced table or graph (vs. basic table) affects patients' self-reported blood pressure measurement (as averaged across two measurements taken at the time of the survey at least 1 minute apart, as per directions of the American Heart Association), and improves interpretations of these two blood pressure readings and of hypothetical blood pressure readings, as well as behavior change intentions.

Aim 3: The investigators will examine whether Aim 2 findings vary by health literacy, age, and SES.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypertension
* Proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wandi Bruine de Bruin, PhD, Principal Investigator — University of Southern California
Locations (1):
- Pitt+Me Patient Registry, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No personal identifiable patient information will be collected.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Pitt+Me Patient Registry at the University of Pittsburgh
Pre-assignment Details: 35 participants were eligible but did not participate in the study
Period: Overall Study
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
Started | 188 | 176 | 178
Completed | 188 | 176 | 178
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph | Total
Number analyzed (Participants) | 188 | 176 | 178 | 542
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.93 (.80) | 50.73 (.89) | 49.46 (.89) | 50.03 (.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 67 | 63 | 185
  Male | 133 | 109 | 115 | 357
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 36 | 41 | 121
  Not Hispanic or Latino | 144 | 140 | 137 | 421
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 2 | 8
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 52 | 40 | 34 | 126
  White | 123 | 132 | 133 | 388
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 4 | 2 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 188 | 176 | 178 | 542
Diagnosed with hypertension or high blood pressure [Count of Participants; unit: Participants] | 188 | 176 | 178 | 542

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Measured Blood Pressure as Instructed (Assessed on Questionnaire)
Description: This outcome measure reflects the number of participants who measured their blood pressure as instructed, after seeing the communication (coded yes=1/no=0), as self-reported on the questionnaire
Time Frame: Questionnaire completed immediately after receiving communication
Measure: Count of Participants; unit: Participants
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
Number analyzed (Participants) | 188 | 176 | 178
Participants | 34 | 47 | 50
Statistical Analysis 1: Comparison: Communication With Basic Table vs Communication With Enhanced Table vs Communication With Enhanced Graph; Enhanced table > Basic table; Test type: Superiority; p = 0.05, Regression, Logistic; Adjusted for respondent characteristics as described in statistical analysis plan; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.00 to 2.79]
Statistical Analysis 2: Comparison: Communication With Basic Table vs Communication With Enhanced Table vs Communication With Enhanced Graph; Enhanced graph > Basic table; Test type: Superiority; p = 0.05, Regression, Logistic; Adjusted for respondent characteristics as described in statistical analysis plan; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.00 to 2.76]

2. Primary Outcome: Number of Participants Who Understood Blood Pressure Readings (Assessed on Questionnaire)
Description: This outcome measure reflects the number of patients who correctly answered two questions about blood pressure readings outside of the normal range, as included on the questionnaire (coded 1=both questions were answered correctly; 0=at least one of the questions was answered incorrectly). The first question asked whether or not blood pressure readings of 132/69 mmHg are considered normal (correct answer=no). The second question asked whether or not blood pressure readings of 142/91 are considered normal (correct answer=no).
Time Frame: Questionnaire completed immediately after receiving communication
Measure: Count of Participants; unit: Participants
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
Number analyzed (Participants) | 188 | 176 | 178
Participants | 166 | 161 | 155
Statistical Analysis 1: Comparison: Communication With Basic Table vs Communication With Enhanced Table vs Communication With Enhanced Graph; Test type: Superiority — Enhanced table > Basic table; p = 0.29, Regression, Logistic; Adjusted for respondent characteristics as described in statistical analysis plan; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.71 to 3.26]
Statistical Analysis 2: Comparison: Communication With Basic Table vs Communication With Enhanced Table vs Communication With Enhanced Graph; Test type: Superiority — Enhanced graph > Basic table; p = 0.90, Regression, Logistic; Adjusted for respondent characteristics as described in statistical analysis plan; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.48 to 1.93]

3. Primary Outcome: Evaluation of Blood Pressure Reading (Provided on Questionnaire)
Description: On a questionnaire, participants indicated their perceptions of how healthy they think their own blood pressure is right now, giving a score on a scale ranging from 1(=very unhealthy) to 5 (=very healthy).
Time Frame: Questionnaire completed immediately after receiving communication
Measure: Mean (Standard Deviation); unit: Score on a scale (1-5)
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
Number analyzed (Participants) | 188 | 176 | 177
Score on a scale (1-5) | 3.04 (.90) | 2.98 (.94) | 2.90 (.89)
Statistical Analysis 1: Comparison: Communication With Basic Table vs Communication With Enhanced Table; Enhanced table > Basic table; Test type: Superiority; p = 0.13, Regression, Linear; Adjusted for respondent characteristics as described in statistical analysis plan; Unst = -0.14, 95% CI 2-sided [-0.32 to 0.04]
Statistical Analysis 2: Comparison: Communication With Basic Table vs Communication With Enhanced Graph; Enhanced graph > Basic table; Test type: Superiority; p = 0.12, Regression, Linear; Adjusted for respondent characteristics as described in statistical analysis plan; Unstandardized B = -0.14, 95% CI 2-sided [-0.32 to 0.04]

4. Primary Outcome: Behavioral Intention Index (Provided on Questionnaire)
Description: On a questionnaire, participants indicated how likely it is that they will try to lose weight, exercise more, take medication as recommended, and talk to their health care provider about improving their blood pressure readings, giving a score on a scale ranging from 1 (=very unlikely) to 5 (=very likely). This outcome measure reflects the average score across items.
Time Frame: Questionnaire completed immediately after receiving communication
Measure: Mean (Standard Deviation); unit: Score on a scale (1-5)
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
Number analyzed (Participants) | 188 | 176 | 178
Score on a scale (1-5) | 3.58 (.83) | 3.45 (.96) | 3.54 (.85)
Statistical Analysis 1: Comparison: Communication With Basic Table vs Communication With Enhanced Table; Test type: Superiority — Enhanced table > Basic table; p = 0.33, Regression, Linear; Unstandardized B = -0.08, 95% CI 2-sided [-0.25 to 0.08]
Statistical Analysis 2: Comparison: Communication With Basic Table vs Communication With Enhanced Graph; Test type: Superiority; p = 0.29, Regression, Linear; Adjusted for respondent characteristics as described in statistical analysis plan; Unstandardized B = -0.09, 95% CI 2-sided [-0.26 to 0.08]

ADVERSE EVENTS:
Time Frame: Participants completed a questionnaire on one day
Arm/Group | Communication With Basic Table | Communication With Enhanced Table | Communication With Enhanced Graph
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/176 | 0/178
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/176 | 0/178
Other Adverse Events (participants affected / at risk) | 0/188 | 0/176 | 0/178

LIMITATIONS AND CAVEATS:
Participants who agree to complete a survey on blood pressure communications are likely not representative of people with hypertension in the general population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04485637/Prot_SAP_ICF_000.pdf